CLINICAL TRIAL: NCT03376386
Title: Adaptive Dose-Escalated Multi-modality Image-guided RadiothErapy (ADMIRE) for Head and Neck Cancer by Twice Re-imaging, Re-delineation and Re-planning During the Course of Radiotherapy
Brief Title: Adaptive Dose-Escalated Multi-modality Image-guided RadiothErapy
Acronym: ADMIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N17ADM
Record Dates: First submitted 2017-09-26; First posted 2017-12-18 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Head and Neck Cancer
Keywords: Adaptive; Image-guided; Radiotherapy; Head and Neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HNSCC receiving (chemo)radiotherapy (Other): Imaging
  Interventions: Radiation: Adaptive dose-Escalated multi-modality image-guided radiotherapy

INTERVENTIONS:
Radiation: Adaptive dose-Escalated multi-modality image-guided radiotherapy — FDG-PET/CT-scan will be used twice during radiotherapy for a mild dose-escalation to the less-responding parts of the tumor. By adapting the radiotherapy plan, these areas will receive 74-78 Gy.

SUMMARY:
Patients with primary head and neck squamous cell carcinoma (HNSCC) planned for treatment with radiotherapy with or without chemotherapy in curative setting will be treated with an adaptive radiotherapy scheme. An FDG-PET/CT scan for re-delineation and re-planning will be made at the end of the second and fourth of week of radiotherapy. The non-responding part of the tumor on FDG-PET will receive a mild dose-escalation. Depending on the metabolic response, the entire tumor will receive 70 Gy or the residual FDG-avid area will receive 74 or 78 Gy.

DETAILED DESCRIPTION:
If there is a complete metabolic response on the FDG-PET after 2 weeks, the entire tumor will receive 70 Gy. If there is a complete metabolic response after 4 weeks of treatment, the residual FDG-avid area will receive 74 Gy. If there also is no complete metabolic response after 4 weeks of treatment, the residual FDG-avid area will receive 78 Gy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic biopsy confirmed squamous cell carcinoma of the oral cavity, HPV-negative oropharynx, HPV-positive oropharynx with a minimum of 10 pack-years, hypopharynx or larynx
* T2-T4
* Scheduled for radiotherapy or radiotherapy with cisplatin or cetuximab

Exclusion Criteria:

* GFR<30
* Other neoplasms with metastases in the previous 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-04-25 (Actual)

PRIMARY OUTCOMES:
the feasibility of the adaptive radiotherapy scheme estimated by the acute toxicities and implementation of the adaptive treatment plans | 1 year
  The feasibility of the adaptive radiotherapy schedule will be rejected in case of:
  Occurrence of intolerable radiation-induced acute toxicities.
the feasibility of the adaptive radiotherapy scheme estimated by the implementation of the adaptive treatment plans | 1 year
  The feasibility of the adaptive radiotherapy schedule will be rejected in case of:
  The inability to implement 80% of the adaptive treatment plans within 2 days from the intended starting day

SECONDARY OUTCOMES:
the toxicity of the adaptive RT scheme | 1 year
  according to the CTCAE v4.0 scoring system
the locoregional tumor control | 1 year
relative response will be calculated for the decrease of the SUV-value | 1 year
  the prognostic value of the FDG-PET/CT-scans

CONTACTS AND LOCATIONS:
Overall Officials: Abrahim Al-Mamgani, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- Netherlands Cancer Institute, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Mamgani A, Kessels R, Gouw ZAR, Navran A, Mohan V, van de Kamer JB, Sonke JJ, Vogel WV. Adaptive FDG-PET/CT guided dose escalation in head and neck squamous cell carcinoma: Late toxicity and oncologic outcomes (The ADMIRE study). Clin Transl Radiat Oncol. 2023 Sep 17;43:100676. doi: 10.1016/j.ctro.2023.100676. eCollection 2023 Nov. PMID 37753461
- [Derived] Gouw ZAR, La Fontaine MD, Vogel WV, van de Kamer JB, Sonke JJ, Al-Mamgani A. Single-Center Prospective Trial Investigating the Feasibility of Serial FDG-PET Guided Adaptive Radiation Therapy for Head and Neck Cancer. Int J Radiat Oncol Biol Phys. 2020 Nov 15;108(4):960-968. doi: 10.1016/j.ijrobp.2020.04.030. Epub 2020 Apr 30. PMID 32361007